CLINICAL TRIAL: NCT07116343
Title: Intrapleural Ropivacaine Infusion in Cardiac Surgery: Randomized Double-blind Controlled Study
Brief Title: Intrapleural Ropivacaine Infusion in Cardiac Surgery
Acronym: IRICS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Saint Petersburg State University, Russia (Other)
Responsible Party: Principal Investigator, Efremov Sergey, Deputy director for science, Saint-Petersburg state university hospital, Saint Petersburg State University, Russia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPBU IRICS study
Record Dates: First submitted 2025-07-29; First posted 2025-08-11 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Cardiac Surgery; Coronary Artery Disease; Valvular Diseases
Keywords: cardiac surgery; quality of recovery; ropivacaine; postoperative analgesia
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrapleural ropivacaine (Experimental)
  Interventions: Drug: Ropivacaine
- Intrapleural placebo (Placebo Comparator)
  Interventions: Drug: 0.9 % NaCl

INTERVENTIONS:
Drug: Ropivacaine — The patient will receive 0.2% ropivacaine (20.0 ml) into the pleural cavity intraoperatively before sternal closure. A continuous infusion of 0.2% ropivacaine will be administered through a microcatheter into the drained pleural cavity, with titration of the infusion rate. The initial infusion rate is set at 10 ml/hour.
  Arms: Intrapleural ropivacaine
Drug: 0.9 % NaCl — The patient will receive 20.0 ml of a 0.9% sodium chloride solution into the pleural cavity intraoperatively, prior to sternal closure. A continuous infusion of 0.9% sodium chloride solution will then be administered through a microcatheter into the drained pleural cavity. The initial infusion rate is set at 10 ml/hour.
  Arms: Intrapleural placebo

SUMMARY:
For many patients, a primary source of postoperative pain following cardiac surgery is the presence of pleural drains, which the surgeon places at the end of the operation and maintains for 1 to 3 days. One promising method of pain management after cardiac surgery is interpleural analgesia, particularly when traditional analgesic methods, such as systemic opioids or epidural anesthesia, may be limited due to the risk of complications. Interpleural analgesia involves the introduction of local anesthetics directly into the pleural cavity through drainage tubes placed after cardiac surgery. This method targets pain receptors in the chest area, providing effective analgesia without significant systemic effects. Several clinical studies have confirmed the safety and efficacy of intrapleural administration of anesthetics after thoracic surgery. The aim of this randomised double-blind placebo controlled study is to test the hypothesis that, in patients after cardiac surgery, the quality of recovery from anesthesia with intrapleural use of ropivacaine is superior to that with a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled cardiac surgery using a standard median sternotomy.
* Planned opening of the pleural cavities.
* Age more than 18 years.
* Signed informed consent to participate in the study.

Exclusion Criteria:

* Contraindications for ropivacaine
* Redo surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2027-09-25 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Quality of recovery after anesthesia (QoR15) questionnaire | 24 hours after surgery
  ranged from 0 to 150 points, where 0 is the worst and 150 is the best.

SECONDARY OUTCOMES:
pO2/FiO2 ratio | 6, 12, 24 hours after surgery
Morphine equvalents, mg/day | 24 hours after surgery
Pain assessed by Visual analog scale | 6, 12, 24, 48 hours
  from 0 to 10 when 0 is worst and 10 is best

OTHER OUTCOMES:
Postoperative complications | at discharge (assessed up to 30 days)
  Composite (myocardial infarction, stroke, delirium, new onset atrial fibrillation, infections)
Hospital mortality | At discharge (assessed up to 6 months)
  Death during hospitalisation
Length of hospitalisation | At discharge (assessed up to 6 months)
  Number of days in hospital during initial hospitalisation
Sternal wound dehiscence | At discharge (assessed up to 6 months)

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - Saint-Petersburg university hospital, Saint Petersburg
  - Primorskiy general hospital #1, Vladivostok

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available by the reasonable request
Supporting Information: Study Protocol, SAP, ICF